CLINICAL TRIAL: NCT03539146
Title: Gastrointestinal Tolerance, Satiation and Sensory Acceptance of Yogurts Containing Dietary Fiber and Coffee Cascara Extract.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Madrid Institute of Rural Development, Agronomy and Food Research (IMIDRA) (Unknown)
Responsible Party: Principal Investigator, Maria Dolores del Castillo, Principal Investigator, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AGL2014-57239-R
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Satiation; Gastrointestinal Tolerance; Organoleptic Appreciation
Keywords: byproducts; functional yogurt; satiety; sensory analysis; sustainable health; novel food ingredient
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Forty volunteers will be randomly distributed in 4 groups that will follow a sequence of treatments according to a balanced latin square design. Treatment days involve the ingestion in acute conditions of a yogurt formulation with a different dietary fiber dose:
  * Cascara control yogurt with 0% dietary fiber.
  * Cascara yogurt with 3% dietary fiber.
  * Cascara yogurt with 7% dietary fiber.
  * Cascara yogurt with 13% dietary fiber.
  Subjects will have a 48h washout period between treatment days to avoid carry-over effects.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control yogurt (Active Comparator): Treatment with a control yogurt with cascara but no dietary fiber.
  Interventions: Other: Control yogurt
- Yogurt with fiber (Experimental): Treatment with yogurts containing cascara and 3%, 7% and 13% of dietary fiber.
  Interventions: Other: Dietary fiber

INTERVENTIONS:
Other: Dietary fiber — Intake of yogurt containing cascara with 0%, 3%, 7%,13% dietary fiber in a crossover design.
  Arms: Yogurt with fiber
Other: Control yogurt — Control yogurt
  Arms: Control yogurt

SUMMARY:
Coffee processing byproducts, such as coffee cascara (outer skin and pulp of the coffee berry), have potential health promoting properties due to the presence of bioactive compounds. Its use as a novel food ingredient is a means of valorizing this fractioin in the elaboration of functional yogurts. The addition of cascara extract in yogurt affects its texture quality. The addition of dietary fiber can help regain the structure of the yogurt's gel. However, secondary gastrointestinal effects associated with acute fiber ingestion must be considered.The aim of this clinical trial is to study the gastrointestinal tolerance, satiation and sensory acceptance of yogurts containing both coffee cascara extract and different doses of commercial soluble dietary fiber.

DETAILED DESCRIPTION:
Forty healthy volunteers will be recruited and distributed into 4 groups following a randomized, blind, crossover design. Yogurt formulations will be administered two hours after the ingestion of a standardized breakfast, as a snack. Yogurt formulations include:

* Control cascara yogurt with 0% dietary fiber.
* Cascara yogurt with 3% dietary fiber.
* Cascara yogurt with 7% dietary fiber.
* Cascara yogurt with 13% dietary fiber.

The study will be conducted in 4 sessions, with at least 48h of washout period between treatment days. Data on gastrointestinal tolerance, satiation and sensory acceptance will be taken on the same day of the treatment using online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.

Exclusion Criteria:

* Food allergies.
* Lactose intolerant.
* Allergic to milk proteins.
* Diagnosed gastrointestinal disease.
* Pregnant, trying to become pregnant or breast feeding.
* Caffeine sensibility.
* Dietary fiber intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tolerance | 2 hours after ingestion
  Self reported gastrointestinal symptoms including bloating, nausea, flatulence, cramping, diarrhea, constipation and rumbling. Severity of symptoms will be measured with a 4-point scale (0= none, 1= mild, 2=moderate, 3= severe).

SECONDARY OUTCOMES:
Satiety | At 0, 15, 60, 115, 125, 150, 180, 210 and 240 minutes after breakfast meal.
  Self reported sensation of satiety, fullness, thirst, desire to eat food and prospective food consumption. Measurements will be conducted using a 100mm visual analogue scale (VAS).
Sensory acceptance | up to 5 minutes (At the moment of eating the yogurt)
  Self reported sensory acceptance of the different yogurts, reporting overall acceptance and liking for the following attributes in a 9 point hedonic scale: appearance, odor, taste and texture.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores del Castillo, PhD, Principal Investigator — Institute of Food Science Research (CIAL-CSIC)
Locations (1):
- Institute of Food Science Research (CIAL-CSIC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No